CLINICAL TRIAL: NCT01995318
Title: Effectiveness of Kinesiotaping in the Treatment of Acute Ankle Sprains
Acronym: KINACAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etimesgut Military Hospital (Other)
Collaborators: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, YAHYA AYHAN ACAR, MD., Etimesgut Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YAcar - 1; EtimesgutMH0001 (Other: EtimesgutMH0001)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2013-11

CONDITIONS: Sprain of Ankle
Keywords: Kinesiotaping
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elastic bandage (Placebo Comparator): Elastic bandage application as one of routine treatment choice of acute ankle sprains.
- Kinesiotaping (Other): Application of anti-edema kinesiotaping
  Interventions: Other: Kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — Application of anti-edema type kinesiotaping to injured ankle.
  Arms: Kinesiotaping

SUMMARY:
Study hypothesis: Kinesiotaping is effective in treatment of acute ankle sprains in emergency department. It enhances Karlsson score more than elastic bandage.

DETAILED DESCRIPTION:
Study design We conducted this prospective, randomized, blinded, clinical study in a tertiary care setting's ED of which had an annual 600000 visits between July 2013 and November 2013.

Selection of participants The patients whom reported an acutely twisted ankle were included in the study. Exclusion criteria were; patients under 18, pregnancy, legally incompetent to take responsibility, fracture at ankle and/or foot, unstable sprains requiring stabilization with cast, 48 hours since injury occurrence, multiple injuries, have neurologic deficit at lower extremities, chronic instability of ankle, had surgical treatment to ankle, knee and hip.

Interventions After signing an informed consent form, eligible subjects were recruited for the study and were randomly assigned to a kinesiotaping group or elastic bandage group. The simple random number table used for randomization. All patients included in the study were given standard therapy which includes rest for 2 days, elevation of the affected ankle from heart level, ice application for 20 minutes 3 times per day for 5 days. The kinesiotaping and elastic bandage were applied for 5 days. . Kinesiotaping group patients received kinesiotaping applications with Kinesio Tex Gold ® tapes. Lymphatic correction was applied depending on the size of ankle with 2 fan cut tapes with light paper-off tension on the medial and lateral aspects of the ankle (3) Both modalities were applied by the same certified researcher.

Pain scores were obtained using numeric pain rating scale (NPRS) from 0 to 10, with 0 analogous to ''no pain'' and 10 equivalent to ''the most severe pain encountered in life''.

Both groups were used also prescribed non-steroidal anti-inflammatory drugs (NSAID- diclofenac sodium 75 mg per oral). After regular use for two days, patients were told to take the additional doses if only they had pain. At the control days, they were questioned whether they used any additional dose.

Active range of motion (ROM) was measured with a standard manual goniometer when patients were seated on a treatment table with the knees fully extended (0°) and the feet hanging off the end of the table.

Follow up measurements were done at 0, 3, 7, and 28 day by a blinded investigator. To provide blinding, in follow ups patients were seen firstly by researcher who applied the kinesiotaping or elastic bandage. Then the application was removed and then the follow-up measurements were done by another researcher who did not know in which group was the patient randomized. After this measurements, primary researcher applied the therapy again. Study was registered to clinicaltrials.org website (ClinicalTrials.gov identifier: NCT01995318).

Sample size was calculated as 28 for each group. (mu (0): 40, mu (1): 48, sigma: 15, two-sided, alpha: 0.05, power of test: 0.80) Outcome measures The primary outcome measure was ankle joint function which was assessed with Karlsson scoring scale at the day seven. This is a statistically validated scoring scale devised by Karlsson and Peterson. From a maximum score of 90, points are given for a series of eight categories assessing the following areas: pain (20 points), swelling (10 points), instability (subjective) (15 points), stiffness (5 points), stair climbing (10 points), running (10 points), work activities (15 points), and the use of a support device (5 points) (4).

Secondary outcome measures were ankle girth (swelling) changes, the difference in NPRS compared with initial presentation and the use of NSAID after 2 days. Ankle girth was defined as the circumferential measurement of the ankle at the level of both malleoli.

Statistically analysis Statistically analysis were performed by SPSS 15.0 packet programme (SPSS Inc, Chicago, IL) Normal distribution was assessed by Kolmogorov-Smirnov test. Differences between groups were analyzed by t-test. For the differences in day 1, 3, and 7 were analyzed with repeated measures variance analysis. Difference between groups in day 28 was analyzed by Mann-Whitney U test. Chi-square test was used to evaluate the difference between two groups in analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients in isolated acute ankle sprains in emergency department.

Exclusion Criteria:

1. Under 18 years
2. Pregnancy
3. Fracture
4. 48 hours after injury
5. Chronic ankle instability
6. Nurologic deficit in lower extremity
7. Multipl trauma patients
8. Ankle, pelvis or knee surgery history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Karlsson score enhancement | 0-3-7 and 28 days after injury

CONTACTS AND LOCATIONS:
Overall Officials: Yahya A ACAR, MD, Study Director — Etimesgut Military Hospital Ankara/Turkey
Locations (1):
- Bagcilar Education and Training Hospital, Istanbul, Turkey (Türkiye)